CLINICAL TRIAL: NCT01239940
Title: RIBS IV (Restenosis Intra-stent of Drug-eluting Stents: Paclitaxel-eluting Balloon vs Everolimus-eluting Stent). A Prospective, Multicenter and Randomized Clinical Trial
Brief Title: RIBS IV (Restenosis Intra-stent of Drug-eluting Stents: Paclitaxel-eluting Balloon vs Everolimus-eluting Stent)
Acronym: RIBS IV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Médica para la Investigación y Desarrollo en el Area Cardiovascular (Other)
Collaborators: Hospital San Carlos, Madrid (Other); B.Braun Surgical SA (Industry); Abbott Medical Devices (Industry)
Responsible Party: Fernando Alfonso, MD, PhD, Hospital Universitario Clinico San Carlos, Madrid. Cardiovascular Institute. Cardiac Department. Interventional Cardiology Unit
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIBS IV
Record Dates: First submitted 2010-11-12; First posted 2010-11-15 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2010-11

CONDITIONS: In-stent Restenosis
Keywords: In-stent restenosis; Drug-eluting balloon; Drug-eluting stent; Angiography; Minimal lumen diameter

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel-eluting balloon (Active Comparator): Paclitaxel-eluting balloon (SeQuent Please, B. Braun)
  Interventions: Device: Coronary angioplasty using the paclitaxel-eluting balloon
- Everolimus-eluting stent (Active Comparator): Everolimus-eluting stent (Xience Prime, Abbott Vascular)
  Interventions: Device: Coronary angioplasty using the Everolimus-eluting stent

INTERVENTIONS:
Device: Coronary angioplasty using the paclitaxel-eluting balloon — Balloon angioplasty
  Arms: Paclitaxel-eluting balloon
Device: Coronary angioplasty using the Everolimus-eluting stent — Stent implantation
  Arms: Everolimus-eluting stent

SUMMARY:
Treatment of patients with drug-eluting stent restenosis remains a challenge. This study will assess which interventional strategy (paclitaxel-eluting balloon vs everolimus-eluting stent) is superior in the treatment of patients suffering from drug-eluting stent restenosis.

DETAILED DESCRIPTION:
Treatment of patients with drug-eluting stent restenosis remains a major clinical and technical challenge. Currently, drug-eluting stents are widely used in the management of these patients. Recently, the value of the paclitaxel-eluting balloon in this clinical setting has been suggested. However, there is only scarce observational data on the value of this new balloon in patients with drug-eluting stent restenosis.

This prospective, multicenter, randomized clinical trial will compare two different interventional strategies (namely, paclitaxel-eluting balloon vs everolimus-eluting stent) in the treatment of patients with drug-eluting stent restenosis.

ELIGIBILITY:
Inclusion Criteria:

PATIENT:

* Age between 20 and 85 years
* Signed informed consent
* Acceptance of late angiographic control (6-9 months)
* Angina and / or objective evidence of ischemia

LESION:

* In-Stent restenosis (> 50% visual) any drug-eluting stent
* Knowledge of prior stent location

Exclusion Criteria:

PATIENT:

* Inclusion in another clinical research protocol
* Women of childbearing age
* Severe associated systemic disease (including renal or liver failure)
* Severe depression of left ventricular ejection fraction (LVEF <25%)
* Disease that affects life expectancy
* Recent myocardial infarction ( <7 days)
* Time of implantation of the previous DES <1 month
* Severe difficulties expected for late angiographic study

LESION:

* Angiographic failure during implementation of initial stent(residual stenosis> 50%)
* Image of large thrombus in-stent (> vessel diameter)
* Tortuosity or Ca + + with very severe difficulties during prior stent deployment
* Vessel diameter <2 mm (visual estimate)
* Restenosis only "outside" the stent (The edge of the stent is not affected)
* Completely occlusive restenosis (100%, TIMI 0)
* Very diffuse restenosis (> 30 mm length)

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Minimal lumen diameter | Late angiographic follow-up (6-9 months)
  Comparison of minimal lumen diameter at late angiographic follow-up (6-9 months) between the 2 treatment strategies (by quantitative coronary angiography)

SECONDARY OUTCOMES:
Combined clinical and angiographic end-points | 6-9 months, 1 year and 3 years
  A) Efficacy outcomes:
  A1) Angiographic: 1) Restenosis rate, 2) % diameter stenosis, 3) acute gain, 4) late loss, 5) net gain A2) Composite of death, myocardial infarction, target vessel revascularization and analysis of individual events
  B) Safety Outcomes: Stent thrombosis, Bleeding episodes.
  C) Pre-specified variables for subgroup analysis (RIBS I)
  D) Stratification (length and edge). Type of stent and eluted drug
  E) Influence of clinical variables and restenosis patterns on outcome

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Alfonso, MD, PhD, Study Director — Hospital San Carlos, Madrid
Locations (25):
- Spain (25):
  - Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña
  - Hospital General Universitario de Alicante, Alicante, Alicante
  - Complejo Hospitalario de Torrecardenas, Almería, Almeria
  - Hospital Universitario Infanta Cristina, Badajoz, Badajoz
  - Hospital Universitari Son Dureta, Palma de Mallorca, Balearic Islands
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Universitari Vall d´Hebron, Barcelona, Barcelona
  - Hospital Clinic de Barcelona, Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Hospital Universitario de La Princesa, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Carlos Haya, Málaga, Malaga
  - Hospital Universitario Virgen de la Victoria, Málaga, Malaga
  - Hospital Provincial de Navarra, Pamplona, Navarre
  - Complejo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Complejo Hospitalario de Toledo, Toledo, Toledo
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza, Zaragoza

REFERENCES:
- [Background] Baz JA, Pinar E, Albarran A, Mauri J; Spanish Society of Cardiology Working Group on Cardiac Catheterization and Interventional Cardiology. Spanish Cardiac Catheterization and Coronary Intervention Registry. 17th official report of the Spanish Society of Cardiology Working Group on Cardiac Catheterization and Interventional Cardiology (1990-2007). Rev Esp Cardiol. 2008 Dec;61(12):1298-314. doi: 10.1016/s1885-5857(09)60057-8. English, Spanish. PMID 19080969
- [Background] Alfonso F, Perez-Vizcayno MJ, Cruz A, Garcia J, Jimenez-Quevedo P, Escaned J, Hernandez R. Treatment of patients with in-stent restenosis. EuroIntervention. 2009 May;5 Suppl D:D70-8. PMID 19736076
- [Background] Pinar E, Albarran A, Baz JA, Mauri J. [Update on interventional cardiology]. Rev Esp Cardiol. 2009 Jan;62 Suppl 1:101-16. doi: 10.1016/s0300-8932(09)70045-4. Spanish. PMID 19174054
- [Background] Daemen J, Wenaweser P, Tsuchida K, Abrecht L, Vaina S, Morger C, Kukreja N, Juni P, Sianos G, Hellige G, van Domburg RT, Hess OM, Boersma E, Meier B, Windecker S, Serruys PW. Early and late coronary stent thrombosis of sirolimus-eluting and paclitaxel-eluting stents in routine clinical practice: data from a large two-institutional cohort study. Lancet. 2007 Feb 24;369(9562):667-78. doi: 10.1016/S0140-6736(07)60314-6. PMID 17321312
- [Background] Hernandez RA, Macaya C, Iniguez A, Alfonso F, Goicolea J, Fernandez-Ortiz A, Zarco P. Midterm outcome of patients with asymptomatic restenosis after coronary balloon angioplasty. J Am Coll Cardiol. 1992 Jun;19(7):1402-9. doi: 10.1016/0735-1097(92)90594-d. PMID 1593031
- [Background] Kimura T, Yokoi H, Nakagawa Y, Tamura T, Kaburagi S, Sawada Y, Sato Y, Yokoi H, Hamasaki N, Nosaka H, et al. Three-year follow-up after implantation of metallic coronary-artery stents. N Engl J Med. 1996 Feb 29;334(9):561-6. doi: 10.1056/NEJM199602293340903. PMID 8569823
- [Background] Lopez-Palop R, Pinar E, Lozano I, Saura D, Pico F, Valdes M. Utility of the fractional flow reserve in the evaluation of angiographically moderate in-stent restenosis. Eur Heart J. 2004 Nov;25(22):2040-7. doi: 10.1016/j.ehj.2004.07.016. PMID 15541841
- [Background] Alfonso F, Perez-Vizcayno MJ, Hernandez R, Goicolea J, Fernandez-Ortiz A, Escaned J, Banuelos C, Fernandez C, Macaya C. Long-term outcome and determinants of event-free survival in patients treated with balloon angioplasty for in-stent restenosis. Am J Cardiol. 1999 Apr 15;83(8):1268-70, A9. doi: 10.1016/s0002-9149(99)00071-5. PMID 10215297
- [Background] Mehran R, Dangas G, Abizaid AS, Mintz GS, Lansky AJ, Satler LF, Pichard AD, Kent KM, Stone GW, Leon MB. Angiographic patterns of in-stent restenosis: classification and implications for long-term outcome. Circulation. 1999 Nov 2;100(18):1872-8. doi: 10.1161/01.cir.100.18.1872. PMID 10545431
- [Background] Alfonso F, Cequier A, Angel J, Marti V, Zueco J, Bethencourt A, Mantilla R, Lopez-Minguez JR, Gomez-Recio M, Moris C, Perez-Vizcayno MJ, Fernandez C, Macaya C, Seabra-Gomes R; Restenosis Intra-stent Balloon angioplasty versus elective Stenting (RIBS) Investigators. Value of the American College of Cardiology/American Heart Association angiographic classification of coronary lesion morphology in patients with in-stent restenosis. Insights from the Restenosis Intra-stent Balloon angioplasty versus elective Stenting (RIBS) randomized trial. Am Heart J. 2006 Mar;151(3):681.e1-681.e9. doi: 10.1016/j.ahj.2005.10.014. PMID 16504631
- [Background] Alfonso F, Suarez A, Perez L, Sabate M, Moreno R, Banuelos C. Intravascular ultrasound in patients with challenging in-stent restenosis: importance of precise stent visualization. J Interv Cardiol. 2006 Apr;19(2):153-9. doi: 10.1111/j.1540-8183.2006.00123.x. PMID 16650244
- [Background] Mehran R, Mintz GS, Popma JJ, Pichard AD, Satler LF, Kent KM, Griffin J, Leon MB. Mechanisms and results of balloon angioplasty for the treatment of in-stent restenosis. Am J Cardiol. 1996 Sep 15;78(6):618-22. doi: 10.1016/s0002-9149(96)00381-5. PMID 8831392
- [Background] Wong SC, Baim DS, Schatz RA, Teirstein PS, King SB 3rd, Curry RC Jr, Heuser RR, Ellis SG, Cleman MW, Overlie P, et al. Immediate results and late outcomes after stent implantation in saphenous vein graft lesions: the multicenter U.S. Palmaz-Schatz stent experience. The Palmaz-Schatz Stent Study Group. J Am Coll Cardiol. 1995 Sep;26(3):704-12. doi: 10.1016/0735-1097(95)00217-r. PMID 7642863
- [Background] Reimers B, Moussa I, Akiyama T, Tucci G, Ferraro M, Martini G, Blengino S, Di Mario C, Colombo A. Long-term clinical follow-up after successful repeat percutaneous intervention for stent restenosis. J Am Coll Cardiol. 1997 Jul;30(1):186-92. doi: 10.1016/s0735-1097(97)00142-3. PMID 9207641
- [Background] Bauters C, Banos JL, Van Belle E, Mc Fadden EP, Lablanche JM, Bertrand ME. Six-month angiographic outcome after successful repeat percutaneous intervention for in-stent restenosis. Circulation. 1998 Feb 3;97(4):318-21. doi: 10.1161/01.cir.97.4.318. PMID 9468204
- [Background] Adamian M, Colombo A, Briguori C, Nishida T, Marsico F, Di Mario C, Albiero R, Moussa I, Moses JW. Cutting balloon angioplasty for the treatment of in-stent restenosis: a matched comparison with rotational atherectomy, additional stent implantation and balloon angioplasty. J Am Coll Cardiol. 2001 Sep;38(3):672-9. doi: 10.1016/s0735-1097(01)01458-9. PMID 11527615
- [Background] Albiero R, Silber S, Di Mario C, Cernigliaro C, Battaglia S, Reimers B, Frasheri A, Klauss V, Auge JM, Rubartelli P, Morice MC, Cremonesi A, Schofer J, Bortone A, Colombo A; RESCUT Investigators. Cutting balloon versus conventional balloon angioplasty for the treatment of in-stent restenosis: results of the restenosis cutting balloon evaluation trial (RESCUT). J Am Coll Cardiol. 2004 Mar 17;43(6):943-9. doi: 10.1016/j.jacc.2003.09.054. PMID 15028348
- [Background] Alfonso F. Should we use the cutting balloon in patients with in-stent restenosis? J Am Coll Cardiol. 2004 Dec 21;44(12):2416; author reply 2417. doi: 10.1016/j.jacc.2004.09.022. No abstract available. PMID 15607412
- [Background] Mehran R, Dangas G, Mintz GS, Waksman R, Abizaid A, Satler LF, Pichard AD, Kent KM, Lansky AJ, Stone GW, Leon MB. Treatment of in-stent restenosis with excimer laser coronary angioplasty versus rotational atherectomy: comparative mechanisms and results. Circulation. 2000 May 30;101(21):2484-9. doi: 10.1161/01.cir.101.21.2484. PMID 10831522
- [Background] Strauss BH, Umans VA, van Suylen RJ, de Feyter PJ, Marco J, Robertson GC, Renkin J, Heyndrickx G, Vuzevski VD, Bosman FT, et al. Directional atherectomy for treatment of restenosis within coronary stents: clinical, angiographic and histologic results. J Am Coll Cardiol. 1992 Dec;20(7):1465-73. doi: 10.1016/0735-1097(92)90438-s. PMID 1360479
- [Background] Sharma SK, Kini A, Mehran R, Lansky A, Kobayashi Y, Marmur JD. Randomized trial of Rotational Atherectomy Versus Balloon Angioplasty for Diffuse In-stent Restenosis (ROSTER). Am Heart J. 2004 Jan;147(1):16-22. doi: 10.1016/j.ahj.2003.07.002. PMID 14691413
- [Background] vom Dahl J, Dietz U, Haager PK, Silber S, Niccoli L, Buettner HJ, Schiele F, Thomas M, Commeau P, Ramsdale DR, Garcia E, Hamm CW, Hoffmann R, Reineke T, Klues HG. Rotational atherectomy does not reduce recurrent in-stent restenosis: results of the angioplasty versus rotational atherectomy for treatment of diffuse in-stent restenosis trial (ARTIST). Circulation. 2002 Feb 5;105(5):583-8. doi: 10.1161/hc0502.103347. PMID 11827923
- [Background] Sabate M, Costa MA, Kozuma K, Kay IP, van der Giessen WJ, Coen VL, Ligthart JM, Serrano P, Levendag PC, Serruys PW. Geographic miss: a cause of treatment failure in radio-oncology applied to intracoronary radiation therapy. Circulation. 2000 May 30;101(21):2467-71. doi: 10.1161/01.cir.101.21.2467. PMID 10831519
- [Background] Waksman R, Ajani AE, White RL, Chan R, Bass B, Pichard AD, Satler LF, Kent KM, Torguson R, Deible R, Pinnow E, Lindsay J. Five-year follow-up after intracoronary gamma radiation therapy for in-stent restenosis. Circulation. 2004 Jan 27;109(3):340-4. doi: 10.1161/01.CIR.0000109488.62415.01. Epub 2004 Jan 19. PMID 14732756
- [Background] Alfonso F, Sabate M. Sirolimus-eluting stents vs brachytherapy for restenosis. JAMA. 2006 Oct 18;296(15):1837-8; author reply 1838. doi: 10.1001/jama.296.15.1837-c. No abstract available. PMID 17047209
- [Background] Holmes DR Jr, Teirstein P, Satler L, Sketch M, O'Malley J, Popma JJ, Kuntz RE, Fitzgerald PJ, Wang H, Caramanica E, Cohen SA; SISR Investigators. Sirolimus-eluting stents vs vascular brachytherapy for in-stent restenosis within bare-metal stents: the SISR randomized trial. JAMA. 2006 Mar 15;295(11):1264-73. doi: 10.1001/jama.295.11.1264. Epub 2006 Mar 12. PMID 16531619
- [Background] Stone GW, Ellis SG, O'Shaughnessy CD, Martin SL, Satler L, McGarry T, Turco MA, Kereiakes DJ, Kelley L, Popma JJ, Russell ME; TAXUS V ISR Investigators. Paclitaxel-eluting stents vs vascular brachytherapy for in-stent restenosis within bare-metal stents: the TAXUS V ISR randomized trial. JAMA. 2006 Mar 15;295(11):1253-63. doi: 10.1001/jama.295.11.1253. Epub 2006 Mar 12. PMID 16531618
- [Background] Moris C, Alfonso F, Lambert JL, Espolita A, Barriales V, Rodriguez V, Barriales R, Cortina A. Stenting for coronary dissection after balloon dilation of in-stent restenosis: stenting a previously stented site. Am Heart J. 1996 Apr;131(4):834-6. doi: 10.1016/s0002-8703(96)90298-7. No abstract available. PMID 8721666
- [Background] Alfonso F, Cequier A, Zueco J, Moris C, Suarez CP, Colman T, Esplugas E, Perez-Vizcayno MJ, Fernandez C, Macaya C. Stenting the stent: initial results and long-term clinical and angiographic outcome of coronary stenting for patients with in-stent restenosis. Am J Cardiol. 2000 Feb 1;85(3):327-32. doi: 10.1016/s0002-9149(99)00741-9. PMID 11078301
- [Background] Mintz GS, Hoffmann R, Mehran R, Pichard AD, Kent KM, Satler LF, Popma JJ, Leon MB. In-stent restenosis: the Washington Hospital Center experience. Am J Cardiol. 1998 Apr 9;81(7A):7E-13E. doi: 10.1016/s0002-9149(98)00190-8. PMID 9551588
- [Background] Shiran A, Mintz GS, Waksman R, Mehran R, Abizaid A, Kent KM, Pichard AD, Satler LF, Popma JJ, Leon MB. Early lumen loss after treatment of in-stent restenosis: an intravascular ultrasound study. Circulation. 1998 Jul 21;98(3):200-3. doi: 10.1161/01.cir.98.3.200. PMID 9697818
- [Background] Alfonso F, Garcia P, Fleites H, Pimentel G, Sabate M, Hernandez R, Escaned J, Banuelos C, Perez-Vizcayno MJ, Moreno R, Macaya C. Repeat stenting for the prevention of the early lumen loss phenomenon in patients with in-stent restenosis. Angiographic and intravascular ultrasound findings of a randomized study. Am Heart J. 2005 Feb;149(2):e1-8. doi: 10.1016/j.ahj.2004.06.022. PMID 15846250
- [Background] Alfonso F, Hernandez C, Perez-Vizcayno MJ, Hernandez R, Fernandez-Ortiz A, Escaned J, Banuelos C, Sabate M, Sanmartin M, Fernandez C, Macaya C. Fate of stent-related side branches after coronary intervention in patients with in-stent restenosis. J Am Coll Cardiol. 2000 Nov 1;36(5):1549-56. doi: 10.1016/s0735-1097(00)00927-x. PMID 11079657
- [Background] Alfonso F, Zueco J, Cequier A, Mantilla R, Bethencourt A, Lopez-Minguez JR, Angel J, Auge JM, Gomez-Recio M, Moris C, Seabra-Gomes R, Perez-Vizcayno MJ, Macaya C; Restenosis Intra-stent: Balloon Angioplasty Versus Elective Stenting (RIBS) Investigators. A randomized comparison of repeat stenting with balloon angioplasty in patients with in-stent restenosis. J Am Coll Cardiol. 2003 Sep 3;42(5):796-805. doi: 10.1016/s0735-1097(03)00852-0. PMID 12957423
- [Background] Alfonso F, Pérez-Vizcayno MJ, Gómez-Recio M, Insa L, Calvo I, Hernández JM, Bullones JA, Hernández R, Escaned J, Macaya C, Gama-Ribeiro V, Leitao-Marques A; Restenosis Intrastent: Balloon Angioplasty Versus Elective Stenting (RIBS) Investigators. Implications of the
- [Background] Alfonso F, Melgares R, Mainar V, Lezaun R, Vazquez N, Tascon J, Pomar F, Cequier A, Angel J, Perez-Vizcayno MJ, Sabate M, Banuelos C, Fernandez C, Garcia JM; Restensois Intra-stent: Ballon angioplasty versus elective Stenting (RIBS) Investigators. Therapeutic implications of in-stent restenosis located at the stent edge. Insights from the restenosis intra-stent balloon angioplasty versus elective stenting (RIBS) randomized trial. Eur Heart J. 2004 Oct;25(20):1829-35. doi: 10.1016/j.ehj.2004.07.019. PMID 15474698
- [Background] Alfonso F, Auge JM, Zueco J, Bethencourt A, Lopez-Minguez JR, Hernandez JM, Bullones JA, Calvo I, Esplugas E, Perez-Vizcayno MJ, Moreno R, Fernandez C, Hernandez R, Gama-Ribeiro V; RIBS Investigators. Long-term results (three to five years) of the Restenosis Intrastent: Balloon angioplasty versus elective Stenting (RIBS) randomized study. J Am Coll Cardiol. 2005 Sep 6;46(5):756-60. doi: 10.1016/j.jacc.2005.05.050. PMID 16139121
- [Background] Alfonso F, Perez-Vizcayno MJ, Hernandez R, Bethencourt A, Marti V, Lopez-Minguez JR, Angel J, Mantilla R, Moris C, Cequier A, Sabate M, Escaned J, Moreno R, Banuelos C, Suarez A, Macaya C; RIBS-II Investigators. A randomized comparison of sirolimus-eluting stent with balloon angioplasty in patients with in-stent restenosis: results of the Restenosis Intrastent: Balloon Angioplasty Versus Elective Sirolimus-Eluting Stenting (RIBS-II) trial. J Am Coll Cardiol. 2006 Jun 6;47(11):2152-60. doi: 10.1016/j.jacc.2005.10.078. PMID 16750678
- [Background] Alfonso F, Perez-Vizcayno MJ, Hernandez R, Bethencourt A, Marti V, Lopez-Minguez JR, Angel J, Iniguez A, Moris C, Cequier A, Sabate M, Escaned J, Jimenez-Quevedo P, Banuelos C, Suarez A, Macaya C; RIBS-II Investigators. Long-term clinical benefit of sirolimus-eluting stents in patients with in-stent restenosis results of the RIBS-II (Restenosis Intra-stent: Balloon angioplasty vs. elective sirolimus-eluting Stenting) study. J Am Coll Cardiol. 2008 Nov 11;52(20):1621-7. doi: 10.1016/j.jacc.2008.08.025. PMID 18992651
- [Background] Alfonso F. Optimal implantation strategies using drug-eluting stents for in-stent restenosis: do we know the answer? Circulation. 2004 Sep 14;110(11):e302. doi: 10.1161/01.CIR.0000141457.02676.FD. No abstract available. PMID 15364823
- [Background] Alfonso F, Perez-Vizcayno MJ, Hernandez R, Fernandez C, Escaned J, Banuelos C, Bethencourt A, Lopez-Minguez JR, Angel J, Cequier A, Sabate M, Moris C, Zueco J, Seabra-Gomes R; Restenosis Intra-Stent: Balloon Angioplasty Versus Elective Stent Implantation (RIBS-I) and Restenosis Intra-Stent: Balloon Angioplasty Versus Elective Sirolimus-Eluting Stenting (RIBS-II) Investigators. Sirolimus-eluting stents versus bare-metal stents in patients with in-stent restenosis: results of a pooled analysis of two randomized studies. Catheter Cardiovasc Interv. 2008 Oct 1;72(4):459-67. doi: 10.1002/ccd.21694. PMID 18814274
- [Background] Kastrati A, Mehilli J, von Beckerath N, Dibra A, Hausleiter J, Pache J, Schuhlen H, Schmitt C, Dirschinger J, Schomig A; ISAR-DESIRE Study Investigators. Sirolimus-eluting stent or paclitaxel-eluting stent vs balloon angioplasty for prevention of recurrences in patients with coronary in-stent restenosis: a randomized controlled trial. JAMA. 2005 Jan 12;293(2):165-71. doi: 10.1001/jama.293.2.165. PMID 15644543
- [Background] Dibra A, Kastrati A, Alfonso F, Seyfarth M, Perez-Vizcayno MJ, Mehilli J, Schomig A. Effectiveness of drug-eluting stents in patients with bare-metal in-stent restenosis: meta-analysis of randomized trials. J Am Coll Cardiol. 2007 Feb 6;49(5):616-23. doi: 10.1016/j.jacc.2006.10.049. Epub 2006 Dec 4. PMID 17276188
- [Background] Alfonso F. Drug-eluting stents and in-stent restenosis. JAMA. 2005 Apr 20;293(15):1855; author reply 1855-6. doi: 10.1001/jama.293.15.1855-a. No abstract available. PMID 15840854
- [Background] Rodriguez AE, Granada JF, Rodriguez-Alemparte M, Vigo CF, Delgado J, Fernandez-Pereira C, Pocovi A, Rodriguez-Granillo AM, Schulz D, Raizner AE, Palacios I, O'Neill W, Kaluza GL, Stone G; ORAR II Investigators. Oral rapamycin after coronary bare-metal stent implantation to prevent restenosis: the Prospective, Randomized Oral Rapamycin in Argentina (ORAR II) Study. J Am Coll Cardiol. 2006 Apr 18;47(8):1522-9. doi: 10.1016/j.jacc.2005.12.052. Epub 2006 Mar 29. PMID 16630986
- [Background] Scheller B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Bohm M, Speck U. Treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. N Engl J Med. 2006 Nov 16;355(20):2113-24. doi: 10.1056/NEJMoa061254. Epub 2006 Nov 13. PMID 17101615
- [Background] Unverdorben M, Vallbracht C, Cremers B, Heuer H, Hengstenberg C, Maikowski C, Werner GS, Antoni D, Kleber FX, Bocksch W, Leschke M, Ackermann H, Boxberger M, Speck U, Degenhardt R, Scheller B. Paclitaxel-coated balloon catheter versus paclitaxel-coated stent for the treatment of coronary in-stent restenosis. Circulation. 2009 Jun 16;119(23):2986-94. doi: 10.1161/CIRCULATIONAHA.108.839282. Epub 2009 Jun 1. PMID 19487593
- [Background] Alfonso F. Paclitaxel-Eluting Balloons for In-Stent Restenosis. Circulation 2010. In press.
- [Background] Lemos PA, van Mieghem CA, Arampatzis CA, Hoye A, Ong AT, McFadden E, Sianos G, van der Giessen WJ, de Feyter PJ, van Domburg RT, Serruys PW. Post-sirolimus-eluting stent restenosis treated with repeat percutaneous intervention: late angiographic and clinical outcomes. Circulation. 2004 Jun 1;109(21):2500-2. doi: 10.1161/01.CIR.0000130173.63105.4E. Epub 2004 May 17. PMID 15148279
- [Background] Cosgrave J, Melzi G, Corbett S, Biondi-Zoccai GG, Babic R, Airoldi F, Chieffo A, Sangiorgi GM, Montorfano M, Michev I, Carlino M, Colombo A. Repeated drug-eluting stent implantation for drug-eluting stent restenosis: the same or a different stent. Am Heart J. 2007 Mar;153(3):354-9. doi: 10.1016/j.ahj.2006.12.009. PMID 17307411
- [Background] Garg S, Smith K, Torguson R, Okabe T, Slottow TL, Steinberg DH, Roy P, Xue Z, Gevorkian N, Satler LF, Kent KM, Suddath WO, Pichard AD, Waksman R. Treatment of drug-eluting stent restenosis with the same versus different drug-eluting stent. Catheter Cardiovasc Interv. 2007 Jul 1;70(1):9-14. doi: 10.1002/ccd.21106. PMID 17580367
- [Background] Whan Lee C, Kim SH, Suh J, Park DW, Lee SH, Kim YH, Hong MK, Kim JJ, Park SW, Park SJ. Long-term clinical outcomes after sirolimus-eluting stent implantation for treatment of restenosis within bare-metal versus drug-eluting stents. Catheter Cardiovasc Interv. 2008 Apr 1;71(5):594-8. doi: 10.1002/ccd.21399. PMID 18311841
- [Background] Steinberg DH, Gaglia MA Jr, Pinto Slottow TL, Roy P, Bonello L, De Labriolle A, Lemesle G, Torguson R, Kineshige K, Xue Z, Suddath WO, Kent KM, Satler LF, Pichard AD, Lindsay J, Waksman R. Outcome differences with the use of drug-eluting stents for the treatment of in-stent restenosis of bare-metal stents versus drug-eluting stents. Am J Cardiol. 2009 Feb 15;103(4):491-5. doi: 10.1016/j.amjcard.2008.09.107. PMID 19195508
- [Background] Gonzalo N, Serruys PW, Okamura T, van Beusekom HM, Garcia-Garcia HM, van Soest G, van der Giessen W, Regar E. Optical coherence tomography patterns of stent restenosis. Am Heart J. 2009 Aug;158(2):284-93. doi: 10.1016/j.ahj.2009.06.004. PMID 19619707
- [Background] Byrne R, Iijima R, Mehilli J, Pache J, Schulz S, Schomig A, Kastrati A. [Treatment of Paclitaxel-eluting stent restenosis with sirolimus-eluting stent implantation: angiographic and clinical outcomes]. Rev Esp Cardiol. 2008 Nov;61(11):1134-9. Spanish. PMID 19000488
- [Background] Colombo A, Latib A. [Treatment of drug-eluting stent restenosis with another drug-eluting stent: do not fail the second time!]. Rev Esp Cardiol. 2008 Nov;61(11):1120-2. No abstract available. Spanish. PMID 19000485
- [Background] ISAR-DESIRE-II. TCT 2009. Abstract.
- [Background] Alfonso F, Garcia J, Perez-Vizcayno MJ, Hernando L, Hernandez R, Escaned J, Jimenez-Quevedo P, Banuelos C, Macaya C. New stent implantation for recurrences after stenting for in-stent restenosis: implications of a third metal layer in human coronary arteries. J Am Coll Cardiol. 2009 Sep 8;54(11):1036-8. doi: 10.1016/j.jacc.2009.04.082. No abstract available. PMID 19729123
- [Background] Stone GW, Midei M, Newman W, Sanz M, Hermiller JB, Williams J, Farhat N, Mahaffey KW, Cutlip DE, Fitzgerald PJ, Sood P, Su X, Lansky AJ; SPIRIT III Investigators. Comparison of an everolimus-eluting stent and a paclitaxel-eluting stent in patients with coronary artery disease: a randomized trial. JAMA. 2008 Apr 23;299(16):1903-13. doi: 10.1001/jama.299.16.1903. PMID 18430909
- [Background] Stone GW, for the SPIRIT IV Investigators. One year clinical results of SPIRIT IV (A Prospective, Randomized Trial Comparing an Everolimus-Eluting Stent and a Paclitaxel-Eluting Stent in Patients with Coronary Artery Disease). Clinical Trials. TCT 2009. San Francisco, USA, Septiembre 2009.
- [Derived] Alfonso F, Perez-Vizcayno MJ, Cuesta J, Garcia Del Blanco B, Garcia-Touchard A, Lopez-Minguez JR, Masotti M, Zueco J, Cequier A, Velazquez M, Moreno R, Mainar V, Dominguez A, Moris C, Molina E, Rivero F, Jimenez-Quevedo P, Gonzalo N, Fernandez-Perez C; RIBS IV Study Investigators (Under the Auspices of the Interventional Cardiology Working Group of the Spanish Society of Cardiology). 3-Year Clinical Follow-Up of the RIBS IV Clinical Trial: A Prospective Randomized Study of Drug-Eluting Balloons Versus Everolimus-Eluting Stents in Patients With In-Stent Restenosis in Coronary Arteries Previously Treated With Drug-Eluting Stents. JACC Cardiovasc Interv. 2018 May 28;11(10):981-991. doi: 10.1016/j.jcin.2018.02.037. PMID 29798776
- [Derived] Alfonso F, Perez-Vizcayno MJ, Garcia Del Blanco B, Garcia-Touchard A, Lopez-Minguez JR, Sabate M, Zueco J, Melgares R, Hernandez R, Moreno R, Dominguez A, Sanchis J, Moris C, Moreu J, Cequier A, Romaguera R, Rivero F, Cuesta J, Gonzalo N, Jimenez-Quevedo P, Cardenas A, Fernandez C; Spanish Society of Cardiology. Usefulness of Drug-Eluting Balloons for Bare-Metal and Drug-Eluting In-Stent Restenosis (from the RIBS IV and V Randomized Trials). Am J Cardiol. 2017 Apr 1;119(7):983-990. doi: 10.1016/j.amjcard.2016.12.006. Epub 2017 Jan 5. PMID 28139220
- [Derived] Alfonso F, Perez-Vizcayno MJ, Garcia Del Blanco B, Garcia-Touchard A, Lopez-Minguez JR, Masotti M, Zueco J, Melgares R, Mainar V, Moreno R, Dominguez A, Sanchis J, Bethencourt A, Moreu J, Cequier A, Marti V, Otaegui I, Bastante T, Gonzalo N, Jimenez-Quevedo P, Cardenas A, Fernandez C; under the auspices of the Interventional Cardiology Working Group of the Spanish Society of Cardiology. Everolimus-Eluting Stents in Patients With Bare-Metal and Drug-Eluting In-Stent Restenosis: Results From a Patient-Level Pooled Analysis of the RIBS IV and V Trials. Circ Cardiovasc Interv. 2016 Jul;9(7):e003479. doi: 10.1161/CIRCINTERVENTIONS.115.003479. PMID 27412868
- [Derived] Alfonso F, Perez-Vizcayno MJ, Cardenas A, Garcia del Blanco B, Garcia-Touchard A, Lopez-Minguez JR, Benedicto A, Masotti M, Zueco J, Iniguez A, Velazquez M, Moreno R, Mainar V, Dominguez A, Pomar F, Melgares R, Rivero F, Jimenez-Quevedo P, Gonzalo N, Fernandez C, Macaya C; RIBS IV Study Investigators (under auspices of Interventional Cardiology Working Group of Spanish Society of Cardiology). A Prospective Randomized Trial of Drug-Eluting Balloons Versus Everolimus-Eluting Stents in Patients With In-Stent Restenosis of Drug-Eluting Stents: The RIBS IV Randomized Clinical Trial. J Am Coll Cardiol. 2015 Jul 7;66(1):23-33. doi: 10.1016/j.jacc.2015.04.063. PMID 26139054
- [Derived] Alfonso F, Perez-Vizcayno MJ, Cardenas A, Garcia Del Blanco B, Garcia-Touchard A, Lopez-Minguez JR, Rivero F, Masotti M, Zueco J, Cequier A, Moris C, Fernandez-Ortiz A, Escaned J, Jimenez-Quevedo P, Gonzalo N, Fernandez C, Macaya C; Restenosis Intra-stent: drug-eluting Balloon vs. everolimus-eluting Stent (RIBS IV) Study Investigators (under the auspices of the Working Group on Interventional Cardiology of the Spanish Society of Cardiology). Rationale and design of the RIBS IV randomised clinical trial (drug-eluting balloons versus everolimus-eluting stents for patients with drug-eluting stent restenosis). EuroIntervention. 2015 Jul;11(3):336-42. doi: 10.4244/EIJY14M09_07. PMID 25244700